CLINICAL TRIAL: NCT00358332
Title: Randomized, Controlled, Dose Escalation Phase I Clinical Trial to Evaluate the Safety and Immunogenicity of WRAIR's AMA-1 Malaria Vaccine (FMP2.1) Adjuvanted in GSKBio's AS02A Vs. Rabies Vaccine in 1-6 Year Old Children in Bandiagara, Mali
Brief Title: Phase I Pediatric FMP2.1/AS02A Trial in Mali
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Walter Reed Army Institute of Research (WRAIR) (U.S. Federal Agency); GlaxoSmithKline (Industry); University of Maryland, Baltimore (Other)
Responsible Party: Director, ORA, HHS/NIAID/DMID
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 05-0146; U19AI065683 (NIH); 2U01AI065683-06 (NIH); GSKBio: Malaria 051 (106874)
Record Dates: First submitted 2006-07-27; First posted 2006-07-31 (Estimated); Results first posted 2009-03-04 (Estimated); Last update posted 2011-10-24 (Estimated); Status verified 2011-10

CONDITIONS: Plasmodium Falciparum Malaria
Keywords: malaria, vaccine, Mali, children
MeSH Terms: conditions — Malaria, Falciparum; Malaria | interventions — Rabies Vaccines

ARMS (3):
- Group 1: FMP2.1/AS02A 10 mcg dose or rabies vaccine. (Experimental): 20 children will be randomized to receive either the 10 mcg dose of FMP2.1/AS02A (n=15) or rabies vaccine (n=5) on study days 0, 30 +/- 7, and 60 +/- 7.
  Interventions: Biological: FMP2.1/AS02A; Biological: Rabies vaccine (RabAvert)
- Group 2: FMP2.1/AS02A 25 mcg dose or rabies vaccine. (Experimental): 40 children will be randomized to receive either the 25 mcg dose of FMP2.1/AS02A (n=30) or rabies vaccine (n=10) on study days 0, 30 +/- 7, and 60 +/- 7.
  Interventions: Biological: FMP2.1/AS02A; Biological: Rabies vaccine (RabAvert)
- Group 3: FMP2.1/AS02A 50 mcg dose or rabies vaccine. (Experimental): 40 children will be randomized to receive either the 50 mcg dose of FMP2.1/AS02A (n=30) or rabies vaccine (n=10) on study days 0, 30 +/- 7, and 60 +/- 7.
  Interventions: Biological: FMP2.1/AS02A; Biological: Rabies vaccine (RabAvert)

INTERVENTIONS:
Biological: FMP2.1/AS02A — FMP2.1 will be reconstituted in AS02A adjuvant. Dosages: 10, 25, or 50 mcg of FMP2.1 or 0.1, 0.25 or 0.5 mL of FMP2.1/AS02A administered by intramuscular injection.
Biological: Rabies vaccine (RabAvert) — RabAvert, white, freeze-dried vaccine for reconstitution with diluent. Dosage: 1.0 mL of rabies vaccine.

SUMMARY:
The purpose of this study is to test the safety and dosages of a malaria vaccine in 100 children, 1-6 years old, in Bandiagara, Mali. The study is testing the safety of the vaccine when it is given to people who are regularly exposed to malaria and it will provide information regarding optimal vaccine dosage. This study will compare 3 injections of different vaccine doses to a rabies vaccine that is already approved. During the study, the child's health will be checked in the clinic and during home visits. Children may participate for about 14 months, and blood will be taken from each child throughout the study. If the child becomes sick from malaria, he/she will be treated. Information from this study may be used to develop a malaria vaccine that will help control the disease.

DETAILED DESCRIPTION:
This study is a randomized, controlled, dose-escalation, phase I trial of the FMP2.1/AS02A malaria vaccine, using rabies vaccine as a control. This study is linked to DMID protocol 07-0003. The primary objective of this study is to evaluate the safety and reactogenicity of FMP2.1/AS02A in children naturally exposed to P. falciparum malaria infection. The secondary objective is to measure the magnitude and duration of antibody response to FMP2.1 by enzyme-linked immunosorbent assay (ELISA). One hundred healthy children aged 1-6 years in Bandiagara, Mali, will be randomized to 1 of 3 possible groups. Twenty subjects will be enrolled in cohort 1 and 40 subjects each in cohorts 2 and 3. Children within each cohort will be randomized in a 3:1 ratio to receive 10, 25 or 50 micrograms of FMP2.1 (in cohorts 1, 2 and 3, respectively) adjuvanted with a proportionate volume of the AS02A, or rabies vaccine. Thus a total of 75 children will receive the malaria vaccine and 25 the rabies vaccine. Immunizations will be given on days 0, 30 and 60 in a staggered fashion, with the first administrations of the 25 and 50 microgram dose levels of FMP2.1 following the first administration of the 10 and 25 microgram dose levels, respectively, by 2-3 weeks. Solicited adverse events will be recorded on the days of immunization and days 1, 2, 3 and 7 after each immunization, and unsolicited adverse events will be recorded for 30 days after each immunization. Children will be followed for 1 year after the last immunization. Sera will be collected for anti-FMP2.1 antibody titers on the days of immunization and 14 days after each immunization as well as 3, 6, 9 and 12 months after the first immunization. Each child will participate in the study for up to 414 days, which includes the screening period. The primary outcome measures include: occurrence of solicited symptoms after each vaccination during a 7-day surveillance period (day of vaccination and days 1, 2, 3 and 7 after vaccination), occurrence of unsolicited symptoms after each vaccination during a 30-day surveillance period (day of vaccination and 30 subsequent days); and occurrence of serious adverse events throughout the study period. The secondary outcome measure is titers and activity of anti-FMP2.1 antibody at each time point where serology samples are analyzed, measured by ELISA.

ELIGIBILITY:
Inclusion Criteria:

* Age 1-6 years inclusive at the time of screening.
* Residing in Bandiagara town.
* Appear to be in generally good health based on clinical and laboratory investigation.
* Separate written informed consent obtained from the parent/guardian before screening and study start, respectively.
* Available to participate in follow-up for the duration of study (14 months).

Exclusion Criteria:

* Previous vaccination with an investigational vaccine or a rabies vaccine.
* Use of a investigational or non-registered drug or vaccine other than the study vaccine(s) within 30 days preceding the first study immunization, or planned use up to 30 days after the third immunization.
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within six months prior to the first immunization. This includes any dose level of oral steroids or inhaled steroids, but not topical steroids.
* Confirmed or suspected immunosuppressive or immunodeficient condition, including human immunodeficiency virus (HIV) infection.
* Confirmed or suspected autoimmune disease.
* History of allergic reactions or anaphylaxis to immunizations or to any vaccine component.
* History of serious allergic reactions to any substance, requiring hospitalization or emergent medical care.
* History of allergy to tetracycline, doxycycline, nickel or Imidazole.
* History of splenectomy.
* Laboratory evidence of liver disease (alanine aminotransferase [ALT] greater than the upper limit of normal of the testing laboratory = 49.6 U/L).
* Laboratory evidence of renal disease (serum creatinine greater than the upper limit of normal of the testing laboratory = 0.5 mg/dL (44.2 micromol/L), or more than trace protein or blood on urine dipstick testing).
* Laboratory evidence of hematologic disease (absolute leukocyte count <5,300/mm^3 or >15,300/mm^3, absolute lymphocyte count <2,300 mm^3, platelet count <133,000/mm^3, or hemoglobin <9.0 g/dL).
* Chronic skin condition that could interfere with vaccine site reactogenicity assessment.
* Administration of immunoglobulins and/or any blood products within the three months preceding the first study immunization or planned administration during the study period.
* Simultaneous participation in any other interventional clinical trial.
* Acute or chronic pulmonary, cardiovascular, hepatic, renal or neurological condition, severe malnutrition, or any other clinical findings that in the opinion of the Principal Investigator (PI) may increase the risk of participating in the study.
* Other condition that in the opinion of the PI would jeopardize the safety or rights of a participant in the trial or would render the participant unable to comply with the protocol.

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2006-11; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Bamako, Malaria Research and Training Center, Bamako, Mali

REFERENCES:
- [Result] Thera MA, Doumbo OK, Coulibaly D, Laurens MB, Kone AK, Guindo AB, Traore K, Sissoko M, Diallo DA, Diarra I, Kouriba B, Daou M, Dolo A, Baby M, Sissoko MS, Sagara I, Niangaly A, Traore I, Olotu A, Godeaux O, Leach A, Dubois MC, Ballou WR, Cohen J, Thompson D, Dube T, Soisson L, Diggs CL, Takala SL, Lyke KE, House B, Lanar DE, Dutta S, Heppner DG, Plowe CV. Safety and immunogenicity of an AMA1 malaria vaccine in Malian children: results of a phase 1 randomized controlled trial. PLoS One. 2010 Feb 4;5(2):e9041. doi: 10.1371/journal.pone.0009041. PMID 20140214

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Parents in Bandiagara Mali were made aware of the study by a radio announcement and voluntarily brought their children to the Bandiagara Malaria Project (BMP) clinic on the campus of the Bandiagara District Hospital in Bandiagara, Mali. The first subject was enrolled on November 3, 2006 and the final subject was enrolled on December 12, 2006.
Groups:
- FMP2.1/AS02A 10 Mcg: Subjects received FMP2.1/AS02A 10 mcg (Falciparum Malaria Protein 2.1 / Adjuvant System 2 of GlaxoSmithKline Biologicals without thimerosal) by intramuscular injection in the deltoid at study days 0, 30 and 60.
- FMP2.1/AS02A 25 Mcg: Subjects received FMP2.1/AS02A 25 mcg (Falciparum Malaria Protein 2.1 / Adjuvant System 2 without thimerosal) by intramuscular injection in the deltoid at study days 0, 30 and 60.
- FMP2.1/AS02A 50 Mcg: Subjects received FMP2.1/AS02A 50 mcg (Falciparum Malaria Protein 2.1 / Adjuvant System 2 without thimerosal) by intramuscular injection in the deltoid at study days 0, 30 and 60.
- RabAvert(R): Subjects received RabAvert(R) rabies vaccine by intramuscular injection in the deltoid at study days 0, 30 and 60.
Period: Overall Study
Arm/Group | FMP2.1/AS02A 10 Mcg | FMP2.1/AS02A 25 Mcg | FMP2.1/AS02A 50 Mcg | RabAvert(R)
Started | 15 | 30 | 30 | 25
Completed | 15 | 27 | 29 | 25
Not Completed | 0 | 3 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FMP2.1/AS02A 10 Mcg | FMP2.1/AS02A 25 Mcg | FMP2.1/AS02A 50 Mcg | RabAvert(R) | Total
Number analyzed (Participants) | 15 | 30 | 30 | 25 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 15 | 30 | 30 | 25 | 100
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 3.5 (1.8) | 3.5 (1.7) | 3.6 (1.7) | 3.2 (1.9) | 3.4 (1.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 15 | 12 | 15 | 49
  Male | 8 | 15 | 18 | 10 | 51
Region of Enrollment [Number; unit: participants]
  Mali | 15 | 30 | 30 | 25 | 100

OUTCOME MEASURES:

1. Primary Outcome: Occurrence of Solicited Systemic Symptoms During a 7-day Surveillance Period (Systematically Collected) Following Vaccinations at Days 0, 30, and 60.
Description: The number of participants reporting drowsiness irritability/fussiness, loss of appetite, vomiting, and feverishness. Participants are counted only once but may have experienced symptoms on multiple occasions.
Time Frame: 7 Days following any vaccination
Population: This outcome includes all enrolled subjects.
Measure: Number; unit: Participants
Arm/Group | FMP2.1/AS02A 10 Mcg | FMP2.1/AS02A 25 Mcg | FMP2.1/AS02A 50 Mcg | RabAvert(R)
Number analyzed (Participants) | 15 | 30 | 30 | 25
Participants
  Drowsiness | 0 | 0 | 0 | 0
  Irritability/Fussiness | 0 | 0 | 0 | 0
  Loss of Appetite | 3 | 0 | 1 | 0
  Vomiting | 2 | 0 | 0 | 0
  Feverishness | 3 | 17 | 16 | 4

2. Primary Outcome: Occurrence of Unsolicited Symptoms During a 30-day Surveillance Period Following Vaccinations at Days 0, 30, and 60.
Description: The number of participants spontaneously reporting any symptom (defined as any Adverse Event considered associated with the product) within 30 days of any vaccination. Participants are counted only once but may have experienced events on multiple occasions.
Time Frame: Day of vaccination and 30 subsequent days.
Population: This outcome includes all enrolled subjects.
Measure: Number; unit: Participants
Arm/Group | FMP2.1/AS02A 10 Mcg | FMP2.1/AS02A 25 Mcg | FMP2.1/AS02A 50 Mcg | RabAvert(R)
Number analyzed (Participants) | 15 | 30 | 30 | 25
Participants | 4 | 7 | 10 | 2

3. Primary Outcome: Number of Subjects Spontaneously Reporting Any Serious Adverse Event.
Description: Any untoward medical occurrence that resulted in death, persistent/significant disability/incapacity, required in-patient hospitalization or prolongation thereof, was life threatening or a congenital anomaly/birth defect in offspring of a study subject; or may have jeopardized the participant or required intervention to prevent one of the outcomes.
Time Frame: 1 year after the last vaccination.
Population: This outcome includes all enrolled subjects.
Measure: Number; unit: Participants
Arm/Group | FMP2.1/AS02A 10 Mcg | FMP2.1/AS02A 25 Mcg | FMP2.1/AS02A 50 Mcg | RabAvert(R)
Number analyzed (Participants) | 15 | 30 | 30 | 25
Participants | 1 | 1 | 0 | 2

4. Secondary Outcome: Anti-FMP2.1 Antibody Titers Measured by ELISA, at Day 0
Description: This outcome is the mean of the log anti-FMP2.1 antibody response measured by ELISA.
Time Frame: Day 0
Population: Participants included are those meeting all eligibility criteria, and who have received at least one immunization with any of the study or control vaccines and for whom immunogenicity data at the indicated time point are available.
Measure: Mean (95% Confidence Interval); unit: log anti-FMP2.1 titer
Arm/Group | FMP2.1/AS02A 10 Mcg | FMP2.1/AS02A 25 Mcg | FMP2.1/AS02A 50 Mcg | RabAvert(R)
Number analyzed (Participants) | 15 | 30 | 30 | 25
log anti-FMP2.1 titer | 2.73 [1.99 to 3.47] | 2.70 [2.22 to 3.17] | 3.04 [2.65 to 3.42] | 2.66 [2.18 to 3.14]

5. Primary Outcome: Occurrence of Solicited Local Symptoms During a 7-day Surveillance Period (Systematically Collected) Following Vaccinations at Days 0, 30, and 60.
Description: The number of participants reporting pain, swelling and erythema. Participants are counted only once but may have experienced symptoms on multiple occasions.
Time Frame: 7 Days following any vaccination
Population: This outcome includes all enrolled subjects.
Measure: Number; unit: Participants
Arm/Group | FMP2.1/AS02A 10 Mcg | FMP2.1/AS02A 25 Mcg | FMP2.1/AS02A 50 Mcg | RabAvert(R)
Number analyzed (Participants) | 15 | 30 | 30 | 25
Participants
  Site Pain | 11 | 27 | 27 | 6
  Swelling | 13 | 28 | 30 | 11
  Erythema | 0 | 0 | 1 | 0

6. Secondary Outcome: Anti-FMP2.1 Antibody Titers Measured by ELISA, at Day 30
Description: This outcome is the mean of the log anti-FMP2.1 antibody response measured by ELISA.
Time Frame: Day 30 +/- 7 days
Population: as for outcome 4
Measure: Mean (95% Confidence Interval); unit: log anti-FMP2.1 titer
Arm/Group | FMP2.1/AS02A 10 Mcg | FMP2.1/AS02A 25 Mcg | FMP2.1/AS02A 50 Mcg | RabAvert(R)
Number analyzed (Participants) | 15 | 30 | 29 | 24
log anti-FMP2.1 titer | 4.09 [3.78 to 4.41] | 4.20 [4.04 to 4.36] | 4.31 [4.18 to 4.44] | 2.57 [2.05 to 3.09]

7. Secondary Outcome: Anti-FMP2.1 Antibody Titers Measured by ELISA, at Day 60
Description: This outcome is the mean of the log anti-FMP2.1 antibody response measured by ELISA.
Time Frame: Day 60 +/- 7 days
Population: as for outcome 4
Measure: Mean (95% Confidence Interval); unit: log anti-FMP2.1 titer
Arm/Group | FMP2.1/AS02A 10 Mcg | FMP2.1/AS02A 25 Mcg | FMP2.1/AS02A 50 Mcg | RabAvert(R)
Number analyzed (Participants) | 15 | 30 | 29 | 24
log anti-FMP2.1 titer | 4.78 [4.61 to 4.96] | 4.98 [4.84 to 5.11] | 4.97 [4.89 to 5.05] | 2.53 [2.03 to 3.03]

8. Secondary Outcome: Anti-FMP2.1 Antibody Titers Measured by ELISA, at Day 90
Description: This outcome is the mean of the log anti-FMP2.1 antibody response measured by ELISA.
Time Frame: Day 90 +/- 10 days
Population: as for outcome 4
Measure: Mean (95% Confidence Interval); unit: log anti-FMP2.1 titer
Arm/Group | FMP2.1/AS02A 10 Mcg | FMP2.1/AS02A 25 Mcg | FMP2.1/AS02A 50 Mcg | RabAvert(R)
Number analyzed (Participants) | 15 | 30 | 29 | 25
log anti-FMP2.1 titer | 4.93 [4.75 to 5.11] | 5.22 [5.06 to 5.37] | 5.05 [4.91 to 5.19] | 2.41 [1.98 to 2.84]

9. Secondary Outcome: Anti-FMP2.1 Antibody Titers Measured by ELISA, at Day 180
Description: This outcome is the mean of the log anti-FMP2.1 antibody response measured by ELISA.
Time Frame: Day 180 +/- 14 days
Population: as for outcome 4
Measure: Mean (95% Confidence Interval); unit: log anti-FMP2.1 titer
Arm/Group | FMP2.1/AS02A 10 Mcg | FMP2.1/AS02A 25 Mcg | FMP2.1/AS02A 50 Mcg | RabAvert(R)
Number analyzed (Participants) | 15 | 29 | 29 | 25
log anti-FMP2.1 titer | 4.53 [4.33 to 4.73] | 4.73 [4.60 to 4.86] | 4.57 [4.42 to 4.72] | 2.15 [1.75 to 2.54]

10. Secondary Outcome: Anti-FMP2.1 Antibody Titers Measured by ELISA, at Day 272.
Description: This outcome is the mean of the log anti-FMP2.1 antibody response measured by ELISA.
Time Frame: Day 272 +/- 14 days
Population: as for outcome 4
Measure: Mean (95% Confidence Interval); unit: log anti-FMP2.1 titer
Arm/Group | FMP2.1/AS02A 10 Mcg | FMP2.1/AS02A 25 Mcg | FMP2.1/AS02A 50 Mcg | RabAvert(R)
Number analyzed (Participants) | 14 | 29 | 29 | 25
log anti-FMP2.1 titer | 4.25 [4.05 to 4.45] | 4.43 [4.29 to 4.58] | 4.51 [4.33 to 4.70] | 2.13 [1.78 to 2.48]

11. Secondary Outcome: Anti-FMP2.1 Antibody Titers Measured by ELISA, at Day 364
Description: This outcome is the mean of the log anti-FMP2.1 antibody response measured by ELISA.
Time Frame: Day 364 +/- 14 days
Population: Participants included are those meeting all eligibility criteria, and who have received at least one immunization with any of the study or control vaccines and for whom immunogenicity data at the indicated time point is available.
Measure: Mean (95% Confidence Interval); unit: log anti-FMP2.1 titer
Arm/Group | FMP2.1/AS02A 10 Mcg | FMP2.1/AS02A 25 Mcg | FMP2.1/AS02A 50 Mcg | RabAvert(R)
Number analyzed (Participants) | 15 | 27 | 29 | 25
log anti-FMP2.1 titer | 4.36 [4.16 to 4.56] | 4.68 [4.46 to 4.91] | 4.42 [4.27 to 4.57] | 2.56 [2.20 to 2.92]

ADVERSE EVENTS:
Time Frame: Solicited symptoms were recorded 7-day surveillance period (day of vaccination and study days 1, 2, 3 and 7) after each dose, and unsolicited AEs were recorded for 30 days after each immunization. SAEs were collected through 1 year post last dose.
Description: The solicited symptoms are reported separately after each vaccination. The occurrence of a solicited symptom on any day(s) at any severity within the 7-day period was considered one event
Arm/Group | FMP2.1/AS02A 10 Mcg | FMP2.1/AS02A 25 Mcg | FMP2.1/AS02A 50 Mcg | RabAvert(R)
Serious Adverse Events (participants affected / at risk) | 1/15 | 1/30 | 0/30 | 2/25
Other Adverse Events (participants affected / at risk) | 15/15 | 30/30 | 30/30 | 25/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FMP2.1/AS02A 10 Mcg (N=15) | FMP2.1/AS02A 25 Mcg (N=30) | FMP2.1/AS02A 50 Mcg (N=30) | RabAvert(R) (N=25)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
White blood cell count increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | FMP2.1/AS02A 10 Mcg (N=15) | FMP2.1/AS02A 25 Mcg (N=30) | FMP2.1/AS02A 50 Mcg (N=30) | RabAvert(R) (N=25)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Splenomegaly (Blood and lymphatic system disorders) | 2 (2) | 2 (2) | 0 (0) | 1 (2)
Tachycardia (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cerumen impaction (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis (Eye disorders) | 2 (8) | 3 (3) | 7 (8) | 5 (5)
Conjunctivitis allergic (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Eye pruritus (Eye disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 12 (13) | 4 (4) | 1 (1)
Aphthous stomatitis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Dental caries (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dental discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 4 (9) | 8 (18) | 10 (14) | 9 (17)
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Gingivitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Oral disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Rectal prolapse (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Salivary hypersecretion (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Tooth loss (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (2) | 5 (5) | 1 (1) | 2 (3)
Asthenia (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pyrexia (Gastrointestinal disorders) | 4 (6) | 9 (13) | 4 (5) | 3 (3)
Jaundice (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Amoebic dysentery (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Bronchiolitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Bronchitis (Infections and infestations) | 6 (14) | 11 (19) | 12 (20) | 11 (18)
Candidiasis (Infections and infestations) | 0 (0) | 2 (3) | 0 (0) | 1 (1)
Ear infection (Infections and infestations) | 5 (6) | 12 (15) | 6 (7) | 10 (11)
Fungal skin infection (Infections and infestations) | 5 (5) | 5 (7) | 9 (9) | 4 (4)
Furuncle (Infections and infestations) | 1 (1) | 2 (3) | 3 (3) | 2 (3)
Gastroenteritis (Infections and infestations) | 1 (1) | 3 (3) | 0 (0) | 3 (3)
Giardiasis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hepatitis A (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Herpetic stomatitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hymenolepiasis (Infections and infestations) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Infection parasitic (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Malaria (Infections and infestations) | 10 (20) | 16 (25) | 21 (28) | 15 (25)
Mumps (Infections and infestations) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Nasopharyngitis (Infections and infestations) | 10 (14) | 13 (22) | 15 (19) | 15 (28)
Oral herpes (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 2 (2) | 3 (3) | 1 (1) | 5 (7)
Pharyngitis (Infections and infestations) | 5 (5) | 4 (6) | 5 (5) | 4 (4)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 4 (4) | 3 (3)
Pyoderma (Infections and infestations) | 5 (8) | 8 (8) | 8 (8) | 10 (10)
Rhinitis (Infections and infestations) | 13 (27) | 17 (30) | 22 (42) | 20 (39)
Skin infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Streptococcal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 6 (7) | 4 (5) | 7 (7) | 6 (7)
Tooth abscess (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Trichomoniasis intestinal (Infections and infestations) | 2 (2) | 3 (4) | 3 (4) | 1 (1)
Typhoid fever (Infections and infestations) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Vulvovaginitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Forearm fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 3 (3) | 6 (6) | 5 (5) | 2 (2)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Cardiac murmur (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
White blood cell count increased (Investigations) | 1 (1) | 0 (0) | 3 (4) | 2 (3)
Pica (Metabolism and nutrition disorders) | 0 (0) | 2 (3) | 0 (0) | 1 (1)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Convulsion (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (3) | 6 (8) | 2 (2) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 11 (15) | 24 (39) | 17 (26) | 18 (34)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 11 (17) | 11 (14) | 9 (13)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Prurigo (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 0 (0) | 1 (1)
Rash papular (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) | 0 (0) | 1 (1)
Skin lesion (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (4) | 2 (2) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting - post dose 1 (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site pain - post dose 1 (General disorders) | 8 (8) | 19 (19) | 16 (16) | 2 (2)
Injection site swelling - post dose 1 (General disorders) | 11 (11) | 12 (12) | 28 (28) | 6 (6)
Pyrexia - post dose 1 (General disorders) | 0 (0) | 9 (9) | 8 (8) | 0 (0)
Anorexia - post dose 1 (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Injection site pain - post dose 2 (General disorders) | 7 (7) | 15 (15) | 19/28 (19) | 4 (4)
Injection site swelling - post dose 2 (General disorders) | 7 (7) | 22 (22) | 22/28 (22) | 4 (4)
Pyrexia - post dose 2 (General disorders) | 2 (2) | 8 (8) | 6/28 (6) | 2 (2)
Anorexia - post dose 2 (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0/28 (0) | 0 (0)
Vomiting - post dose 3 (Gastrointestinal disorders) | 1/14 (1) | 0/27 (0) | 0/27 (0) | 0/23 (0)
Injection site pain - post dose 3 (General disorders) | 3/14 (3) | 12/27 (12) | 16/27 (16) | 1/23 (1)
Injection site swelling - - post dose 3 (General disorders) | 10/14 (10) | 16/27 (16) | 23/27 (23) | 3/23 (3)
Pyrexia - post dose 3 (General disorders) | 2/14 (2) | 5/27 (5) | 7/27 (7) | 4/23 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less